CLINICAL TRIAL: NCT05655442
Title: Effect of Early vs Delayed Arthroscopic Partial Meniscectomy on the Knee Function of Patients With Degenerative Meniscus Lesions
Brief Title: Arthroscopic Partial Meniscectomy Time Window
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enough participants recruited
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SZlesions
Record Dates: First submitted 2022-12-07; First posted 2022-12-19 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Meniscus Lesion

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early APM (Experimental): early APM within 3 and 6 month knee pain symptoms
  Interventions: Procedure: early APM
- delayed APM (Active Comparator): delayed APM within 6 and 12 month knee pain symptoms
  Interventions: Procedure: delayed APM

INTERVENTIONS:
Procedure: early APM — early APM within 3 and 6 month knee pain symptoms
  Arms: early APM
Procedure: delayed APM — delayed APM within 6 and 12 month knee pain symptoms
  Arms: delayed APM

SUMMARY:
The purpose was to assess knee function outcomes between early arthroscopic partial meniscectomy(APM) and delayed APM for patients with degenerative meniscus lesions(DMLs)

DETAILED DESCRIPTION:
Whether early APM surgery or delayed APM surgery will more benefit for patients with DMLs. The study was to determine the early APM vs delayed APM effect on knee function outcomes for patients with DMLs for 1 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* • Clinical diagnosis of degenerative meniscus lesions based on knee MRI

Exclusion Criteria:

* • Must be able to have no acute knee injury such as car crash or acute sports injury;

  * Must be able to have no knee surgeries history;
  * Must be able to have no rheumatoid arthritis or serious knee osteoarthritis with deformity;
  * Must be able to have no contraindications to MRI;
  * Must be able to have no severe cardiopulmonary disease;
  * Must be able to have no musculoskeletal or neuromuscular impairments ;
  * Must be able to have good visual, hearing, or cognitive;

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-12 (Actual); Primary Completion 2023-07-05 (Estimated); Study Completion 2023-08-28 (Estimated)

PRIMARY OUTCOMES:
the Knee Injury and Osteoarthritis Outcome Score (KOOS) change | change from baseline up to 12 months
  The Knee injury and Osteoarthritis Outcome Score (KOOS) holds five subscales including: Pain (9 items); other Symptoms (7 items); Activities of Daily Living (ADL, 17 items); Sport and Recreation function (Sport/Rec, 5 items); and knee-related Quality of Life (QoL, 4 items). Each subscale is scored separately from zero (extreme knee problems) to 100 (no knee problems)
International Knee Documentation Committee Subjective Knee Evaluation Form (IKDC Score) change | change from baseline up to 12 months
  The International Knee Documentation Committee Subjective Knee Evaluation Form (IKDC) score questionnaire contains 18 items (7 items for symptoms, 1 item for sport activity, 9 items for daily activities, and 1 item for current knee function.) The total score is transformed to a value on a scale of 0 to 100, with 100 representing the highest knee function and 0 is the worst.
Kellgren-Lawrence (K/L) grade change | change from baseline up to 12 months
  Kellgren-Lawrence (K/L) grade via X ray
the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) change | change from baseline up to 12 months
  Te WOMAC is a self assessed health status scale for patients consisting of 24 items in three subscales of pain (5 items), stiffness (2 items), and physical function (17 items). All items are scored from 0 (asymptomatic) to 4 (very severe), and the total score ranges from 0 to 96, with higher scores indicating more severe symptoms

SECONDARY OUTCOMES:
KOOS pain score change | change from baseline up to 12 months
  The minimum is 0 points, the maximum is 4 points, from extreme knee problems to no knee problems. After the score of each part is calculated separately, it is converted into a percentage score by the conversion formula.
KOOS symptoms score change | change from baseline up to 12 months
  The minimum is 0 points, the maximum is 4 points, from extreme knee problems to no knee problems. After the score of each part is calculated separately, it is converted into a percentage score by the conversion formula.
KOOS activities of daily living score change | change from baseline up to 12 months
  The minimum is 0 points, the maximum is 4 points, from extreme knee problems to no knee problems. After the score of each part is calculated separately, it is converted into a percentage score by the conversion formula.
KOOS function in sport and recreation score change | change from baseline up to 12 months
  The minimum is 0 points, the maximum is 4 points, from extreme knee problems to no knee problems. After the score of each part is calculated separately, it is converted into a percentage score by the conversion formula.
KOOS knee related quality of life score change | change from baseline up to 12 months
  The minimum is 0 points, the maximum is 4 points, from extreme knee problems to no knee problems. After the score of each part is calculated separately, it is converted into a percentage score by the conversion formula.

CONTACTS AND LOCATIONS:
Overall Officials: Hongyu Wang, Doctor, Principal Investigator — Shenzhen People's Hospital

IPD SHARING:
Plan to Share IPD: No